CLINICAL TRIAL: NCT06713642
Title: SPOTFIRE ST TITUS STUDY: Provider Identified Target Populations, Implementation, Test Performance, Potential Utility, and Satisfaction of SPOTFIRE ST in the Urgent Care
Brief Title: SPOTFIRE Sore Throat (ST) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: BioMérieux (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-1569; Protocol Approved: 10/11/24 (Other: UW Madison); A534265 (Other: UW Madison); BFD-RST-23-010 (Other: Sponsor Protocol ID)
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Pharyngitis, Infective
Keywords: diagnostic test
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Eligible SPOTFIRE ST Participants (Experimental): A maximum of 200 patients, representing the top 3-4 patient groups that were identified as benefitting most from a SPOTFIRE ST test through the provider survey, presenting at the Urgent Care facilities, will be enrolled.
  Interventions: Device: SPOTFIRE ST System

INTERVENTIONS:
Device: SPOTFIRE ST System — Polymerase chain reaction (PCR) test that identifies up to 13 different viral and bacterial pathogens in about 20 Minutes
  Other Names: SPOTFIRE ST

SUMMARY:
The purpose of this study is to evaluate where urgent care (UC) clinicians see the most benefit for a novel, point of care pharyngitis test, SPOTFIRE ST, and describe its performance, potential clinical utility, and satisfaction of providers and patients with this novel test. Up to 200 participants will be on study for up to approximately 25 minutes.

DETAILED DESCRIPTION:
The broader study is separated into three specific aims.

AIM 1. Evaluate which specific patient populations UC providers see the most need and benefit from SPOTFIRE ST, a multiplex point of care pharyngitis test.

AIM 2. Evaluate the performance and effects of test results associated with important clinical outcomes (e.g., prescriptions, additional testing, disposition and follow-up) for patients in the top 3-4 high-risk subpopulations identified by providers in Specific AIM 1.

AIM 3. Evaluate patient and provider satisfaction and future use opportunities of the SPOTFIRE ST Panel testing platform in the clinical pathway for evaluating patients with pharyngitis in UC centers.

AIMS 2-3 are registered to this ClinicalTrials.gov record.

ELIGIBILITY:
Inclusion Criteria:

* Illness onset in the last 7 days, AND:

  * Ages 1-2 (12-35 months old) with fever or
  * Ages 3-17 with sore throat or
  * Any age with immunocompromising conditions or is on immunocompromising medications with sore throat or
  * Any age with comorbidities (e.g., respiratory, cardiovascular, metabolic, renal, etc.) with sore throat

Exclusion Criteria:

* Anatomic anomalies that would prohibit safely collecting a pharyngeal swab specimen
* Symptom onset more than 7 days prior to arrival at urgent care
* Patient is already on an antiviral medication or an antibiotic medication
* Previous participation in the study
* Unable to read and understand or refusal to sign the appropriate informed consent/assent forms
* Refusal to provide their demographics, household information

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Aim 2 Clinical Outcome: Summary of test results | up to 20 minutes
  SPOTFIRE ST results by count.
Aim 2 Clinical Outcome: Number of Participants with follow up testing | up to 3 weeks
  Data collected via electronic medical record review 3 weeks post study visit.
Aim 2 Clinical Outcome: Summary of Resultant Prescriptions | up to 3 weeks
  SPOTFIRE ST resultant prescriptions by count. Data collected via electronic medical record review 3 weeks post study visit.
Aim 3: Participant Satisfaction Survey | emailed after SPOTFIRE testing, survey data collected from all participants through the end of the study (up to 4 months)
  Participant Satisfaction will be measured using a self-report survey scored from 0-10 where higher scores indicate increased satisfaction with the testing experience.
Aim 3: Provider Satisfaction Survey | emailed after SPOTFIRE testing, survey data collected from all participants through the end of the study (up to 4 months)
  Provider Satisfaction will be measured using a self-report survey scored from 0-10 where higher scores indicate increased satisfaction with the testing experience.
Aim 3: Provider Utility Survey | emailed after SPOTFIRE testing, survey data collected from all participants through the end of the study (up to 4 months)
  Providers will be surveyed to learn how they might use the SPOTFIRE test in the future. Survey responses will be ranked and reported by response rate.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Lepak, MD, Principal Investigator — UW School of Medicine and Public Health
Locations (1):
- UW Health Urgent Care Centers, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No